CLINICAL TRIAL: NCT03230513
Title: Comparison of Home-Based Modified Self-Epley Manoeuvre and Brandt-Daroff Exercise on the Posterior Canal Benign Paroxysmal Positional Vertigo Symptoms: A Randomized Single-Blind Controlled Trial
Brief Title: Comparison of Home-Based Exercise on the Posterior Canal Benign Paroxysmal Positional Vertigo Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MREC ID NO: 20155-1337
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: vertigo; benign paroxysmal positional vertigo; particle repositioning manoeuvre
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo

STUDY DESIGN:
Intervention Model Description: Participants were assigned to either the SEM group (written as "Group A") or the BDE group (written as "Group B") throughout the duration of the study.
Who Masked: Investigator
Masking Description: The Primary Investigator (PI) was blinded as to the exercise type that the patient had learned and used and evaluates all the outcomes of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self Epley Manoeuvre (Active Comparator): Self Epley Manoeuvre.
  Interventions: Other: Self Epley Manoeuvre
- Brandt-Daroff Exercise (Active Comparator): Brandt-Daroff Exercise.
  Interventions: Other: Brandt-Daroff Exercise

INTERVENTIONS:
Other: Self Epley Manoeuvre — The patient has to position himself long sitting on the bed, then turn his head 45 degrees to the problematic side. When in this head position, he will rapidly lie himself supine with a pillow under his shoulders. He then turns his head 90 degrees to the opposite direction followed by turning of his body to the same side before returning to a sitting position at the edge of the bed. Each position should be kept for 30 seconds each, and the patient is required to perform 3 cycles of this manoeuvre just prior to going to bed daily for 2 weeks.
  Other Names: SEM
  Arms: Self Epley Manoeuvre
Other: Brandt-Daroff Exercise — The patient has to sit at the edge of the bed, turn his head laterally 45 degrees to one side and move rapidly into the side lying position, keeping his head in the same position. He then returns upright and turns his head to the opposite direction and the same movement is repeated on the other side. Each position is held for at least 30 seconds and the patient is required to perform it for 5 repetitions, three times a day, daily for 2 weeks duration.
  Other Names: BDE
  Arms: Brandt-Daroff Exercise

SUMMARY:
Benign paroxysmal positional vertigo (BPPV) is the most common vestibular disorder in adults and the treatment of choice is by particle repositioning manoeuvres (PRM). This study aims to compare the treatment efficacy of two home-based exercises, self-Epley manoeuvre (SEM) and Brandt-Daroff exercise (BDE) in patients with posterior canal BPPV based on vertigo resolution, reduction of vertigo intensity, the Dizziness Handicap Inventory scores and the conversion of a positive to negative Dix-Hallpike test.

DETAILED DESCRIPTION:
Study Objective:

To compare the efficacy of the self-Epley manoeuvre to the Brandt-Daroff exercise in resolving vertigo symptoms in patients with unilateral posterior canal BPPV.

Study Design:

Single-blind randomized controlled study

Sample Size:

Fifty patients were recruited in the study and were divided with 25 patients in each treatment arm.

Study Method:

Patients who satisfy the inclusion criteria and have given informed consent were randomized into the 2 treatment groups. A dedicated physiotherapist will demonstrate the selected exercise (either SEM or BDE) and observed the patient performing the exercise twice to ensure the ability of the patient to perform it correctly at home. A diary was provided for the patients to chart the therapy sessions performed at home as well as a pamphlet with simple illustrated instructions of the chosen exercise. The patients were asked to perform the home-based exercise for 2 weeks.

Primary Outcome Measure

- Resolution of vertigo symptoms in patients with unilateral posterior canal BPPV.

Secondary Outcome Measures

* Vertigo resolution at 1 and 6 months;
* The conversion of positive to negative Dix-Hallpike test between both groups after 1 month;
* Vertigo intensity in unresolved vertigo patients at 1 & 6 months;
* The Dizziness Handicap Inventory between both groups at 1 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* patients who have had symptoms of vertigo for at least 1 week duration,
* patients with a documented positive Dix-Hallpike test on referral,
* patients with intact cognitive function and had the ability to communicate and understand instructions to perform a home-based exercise.

Exclusion Criteria:

* patients with history of prior ear surgery,
* patients with orthopaedic or connective tissue disorder that impairs functional neck or trunk range of motion,
* patients with a significant neurological disorder or spinal cord damage, and
* patients who have been prescribed with home-based exercises for BPPV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Vertigo resolution | Assessed at 1 month and 6 months following initiation of home-based exercise.
  Present or absent

SECONDARY OUTCOMES:
Conversion of a positive to negative Dix-Hallpike test | Assessed at 1 month following initiation of home-based exercise.
  Positive or negative
Vertigo intensity | Assessed on first assessment during recruitment, at 1 month and 6 months following initiation of home-based exercise.
  Patients were asked to rate the average severity or intensity of the vertigo episode in the previous one week based on a 1-to-5 Likert scale, with a scale of 5 implying the most intense or severe.
Dizziness Handicap Inventory | Assessed on first assessment during recruitment, at 1 month and 6 months following initiation of home-based exercise.
  A 25 item questionnaire that encompasses 3 domains which are functional, physical and emotional. The scores are summed with maximum score of 100 and the higher the score, the greater the perceived handicap.

CONTACTS AND LOCATIONS:
Overall Officials: Mazlina Mazlan, MBBS, MRM, Study Chair — University of Malaya; Nor Hanim Mohamad Hanapi, MBBS, Principal Investigator — University of Malaya

IPD SHARING:
Plan to Share IPD: Undecided